CLINICAL TRIAL: NCT00655733
Title: Double-blind, Randomized, Multicenter, Placebo-controlled Phase II Study of Efficacy and Safety of HMPL-004 in Subjects With Active Moderate Crohn's Disease
Brief Title: Phase II Study of HMPL-004 in Subjects With Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200500401
Record Dates: First submitted 2008-04-06; First posted 2008-04-10 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2018-08

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Andrographis paniculata extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HMPL-004 (Experimental): Subjects who fulfilled all entry criteria and randomized HMPL-004 arm will receive HMPL-004 400 mg 3 times daily 3 times daily for 56 days (8 weeks) with a 28-day (4-week) follow-up.
  Interventions: Drug: HMPL-004
- Placebo (Placebo Comparator): Subjects who fulfilled all entry criteria and randomized Placebo arm will receive matching placebo 400 mg 3 times daily 3 times daily for 56 days (8 weeks) with a 28-day (4-week) follow-up.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HMPL-004 — HMPL-004 1200 mg/d
  Other Names: Chuan xinlian
  Arms: HMPL-004
Drug: Placebo — Placebo 1200 mg/d
  Arms: Placebo

SUMMARY:
A double blind, randomized, multi-center, placebo-controlled study to evaluate the efficacy and safety of HMPL-004 in patients with active moderate Crohn's Disease.

DETAILED DESCRIPTION:
This was a double-blind, randomized, multicenter, placebo-controlled study evaluating the efficacy and safety of oral HMPL-004 in subjects with active moderate Crohn's disease (CD) - Crohn's Disease Activity Index (CDAI) 220 to 400 - on stable doses of CD medications who had not received anti-tumor necrosis factor alpha (anti-TNF-α) for at least 3 months prior to start of treatment. HMPL-004 (or placebo) was added to the subject's existing CD medications. Subjects were observed for an 8-week treatment period and a subsequent 4-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Have active confirmed Crohn's Disease (confirmed radiographically, endoscopic, or histologically), with a CDAI of 220-400 at baseline screen

Exclusion Criteria:

* They have received anti-TNF-α antibody within 3 months of starting study medication, or cyclosporine, tacrolimus, thalidomide or mycophenolate mofetil within 2 months of starting study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rongjun Liu, MD, Study Director — Hutchison Medipharma Limited

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HMPL-004 | Placebo
Started | 51 | 50
Completed | 44 | 42
Not Completed | 7 | 8
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HMPL-004 | Placebo | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 44 | 93
  >=65 years | 2 | 6 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (13.4) | 46.5 (14.2) | 44.4 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 23 | 21 | 44
Region of Enrollment [Number; unit: participants]
  United States | 38 | 35 | 73
  Ukraine | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: CDAI Clinical Response -100 at Week 8
Description: Percentage of subjects with CDAI clinical response -100 at Week 8 based on ITT population using the WOCF method to impute missing CDAI scores at Week 8.
  Clinical response -100 was defined as CDAI score decrease of ≥100 points from baseline in subjects who had no change in concomitant medications for Crohn's disease except for steroids, which could be tapered after Week 8.
  The CDAI consists of eight variables, including Liquid or very soft stools, Abdominal pain, General well-being, Features of extra-intestinal disease, Oplates for diarrhea, Abdominal mass, Hematocrit and Body weight below standard, each weighted according to its ability to be predictive of disease activity. The total score ranges from 0 to over 600 with higher scores indicating higher disease activity or worse outcome.
Time Frame: 8 weeks
Population: Intention-to-treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | HMPL-004 | Placebo
Number analyzed (Participants) | 51 | 50
Participants | 19 | 11

2. Secondary Outcome: Clinical Response -100 at Weeks 4
Description: Percentage of subjects with CDAI clinical response -100 at Week 4 based on ITT population using the WOCF method to impute missing CDAI scores at Week 4.
  Clinical response -100 was defined as CDAI score decrease of ≥100 points from baseline in subjects who had no change in concomitant medications for Crohn's disease except for steroids, which could be tapered after Week 8.
  The CDAI consists of eight variables, including Liquid or very soft stools, Abdominal pain, General well-being, Features of extra-intestinal disease, Oplates for diarrhea, Abdominal mass, Hematocrit and Body weight below standard, each weighted according to its ability to be predictive of disease activity. The total score ranges from 0 to over 600 with higher scores indicating higher disease activity or worse outcome.
Time Frame: 4 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | HMPL-004 | Placebo
Number analyzed (Participants) | 51 | 50
Participants | 15 | 13

3. Secondary Outcome: Clinical Response -100 at Weeks 12
Description: Percentage of subjects with CDAI clinical response -100 at Week 12 based on ITT population using the WOCF method to impute missing CDAI scores at Week 12.
  Clinical response -100 was defined as CDAI score decrease of ≥100 points from baseline in subjects who had no change in concomitant medications for Crohn's disease except for steroids, which could be tapered after Week 8.
  The CDAI consists of eight variables, including Liquid or very soft stools, Abdominal pain, General well-being, Features of extra-intestinal disease, Oplates for diarrhea, Abdominal mass, Hematocrit and Body weight below standard, each weighted according to its ability to be predictive of disease activity. The total score ranges from 0 to over 600 with higher scores indicating higher disease activity or worse outcome.
Time Frame: 12 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | HMPL-004 | Placebo
Number analyzed (Participants) | 51 | 50
Participants | 17 | 11

4. Secondary Outcome: Remission at Week 4
Description: Percentage of subjects achieving remission (CDAI<150) at week 4. Remission was defined as CDAI score <150 in subjects who had no change in concomitant medications for Crohn's disease except for steroids, which could be tapered after Week 8.
  The CDAI consists of eight variables, including Liquid or very soft stools, Abdominal pain, General well-being, Features of extra-intestinal disease, Oplates for diarrhea, Abdominal mass, Hematocrit and Body weight below standard, each weighted according to its ability to be predictive of disease activity. The total score ranges from 0 to over 600 with higher scores indicating higher disease activity or worse outcome.
Time Frame: 4 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | HMPL-004 | Placebo
Number analyzed (Participants) | 51 | 50
Participants | 8 | 8

5. Secondary Outcome: Remission at Week 8
Description: Percentage of subjects achieving remission (CDAI<150) at week 8. Remission was defined as CDAI score <150 in subjects who had no change in concomitant medications for Crohn's disease except for steroids, which could be tapered after Week 8.
  The CDAI consists of eight variables, including Liquid or very soft stools, Abdominal pain, General well-being, Features of extra-intestinal disease, Oplates for diarrhea, Abdominal mass, Hematocrit and Body weight below standard, each weighted according to its ability to be predictive of disease activity. The total score ranges from 0 to over 600 with higher scores indicating higher disease activity or worse outcome.
Time Frame: 8 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | HMPL-004 | Placebo
Number analyzed (Participants) | 51 | 50
Participants | 15 | 7

6. Secondary Outcome: Remission at Week 12
Description: Percentage of subjects achieving remission (CDAI<150) at week 12. Remission was defined as CDAI score <150 in subjects who had no change in concomitant medications for Crohn's disease except for steroids, which could be tapered after Week 8.
  The CDAI consists of eight variables, including Liquid or very soft stools, Abdominal pain, General well-being, Features of extra-intestinal disease, Oplates for diarrhea, Abdominal mass, Hematocrit and Body weight below standard, each weighted according to its ability to be predictive of disease activity. The total score ranges from 0 to over 600 with higher scores indicating higher disease activity or worse outcome.
Time Frame: 12 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | HMPL-004 | Placebo
Number analyzed (Participants) | 51 | 50
Participants | 10 | 7

7. Secondary Outcome: Clinical Response -70 at Week 4
Description: Percentage of patients achieving clinical response -70 at Week 4 (WOCF). Clinical response -70 was defined as CDAI score decrease of ≥70 points from baseline in subjects who had no change in concomitant medications for Crohn's disease except for steroids, which could be tapered after Week 8.
  The CDAI consists of eight variables, including Liquid or very soft stools, Abdominal pain, General well-being, Features of extra-intestinal disease, Oplates for diarrhea, Abdominal mass, Hematocrit and Body weight below standard, each weighted according to its ability to be predictive of disease activity. The total score ranges from 0 to over 600 with higher scores indicating higher disease activity or worse outcome.
Time Frame: 4 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | HMPL-004 | Placebo
Number analyzed (Participants) | 51 | 50
Participants | 20 | 19

8. Secondary Outcome: Clinical Response -70 at Week 8
Description: Percentage of patients achieving clinical response -70 at Week 8 (WOCF). Clinical response -70 was defined as CDAI score decrease of ≥70 points from baseline in subjects who had no change in concomitant medications for Crohn's disease except for steroids, which could be tapered after Week 8.
  The CDAI consists of eight variables, including Liquid or very soft stools, Abdominal pain, General well-being, Features of extra-intestinal disease, Oplates for diarrhea, Abdominal mass, Hematocrit and Body weight below standard, each weighted according to its ability to be predictive of disease activity. The total score ranges from 0 to over 600 with higher scores indicating higher disease activity or worse outcome.
Time Frame: 8 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | HMPL-004 | Placebo
Number analyzed (Participants) | 51 | 50
Participants | 25 | 16

9. Secondary Outcome: Clinical Response -70 at Week 12
Description: Percentage of patients achieving clinical response -70 at Week 12 (WOCF). Clinical response -70 was defined as CDAI score decrease of ≥70 points from baseline in subjects who had no change in concomitant medications for Crohn's disease except for steroids, which could be tapered after Week 8.
  The CDAI consists of eight variables, including Liquid or very soft stools, Abdominal pain, General well-being, Features of extra-intestinal disease, Oplates for diarrhea, Abdominal mass, Hematocrit and Body weight below standard, each weighted according to its ability to be predictive of disease activity. The total score ranges from 0 to over 600 with higher scores indicating higher disease activity or worse outcome.
Time Frame: 12 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | HMPL-004 | Placebo
Number analyzed (Participants) | 51 | 50
Participants | 20 | 18

10. Secondary Outcome: Complete Remission at Week 4
Description: Percentage of subjects achieving complete remission (clinical response -100 plus CDAI<150) at week 4 (WOCF).
  Complete remission was defined as CDAI score decrease of ≥100 points from baseline and CDAI score <150 in subjects who had no change in concomitant medications for Crohn's disease except for steroids, which could be tapered after Week 8.
  The CDAI consists of eight variables, including Liquid or very soft stools, Abdominal pain, General well-being, Features of extra-intestinal disease, Oplates for diarrhea, Abdominal mass, Hematocrit and Body weight below standard, each weighted according to its ability to be predictive of disease activity. The total score ranges from 0 to over 600 with higher scores indicating higher disease activity or worse outcome.
Time Frame: 4 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | HMPL-004 | Placebo
Number analyzed (Participants) | 51 | 50
Participants | 8 | 8

11. Secondary Outcome: Complete Remission at Week 8
Description: Percentage of subjects achieving complete remission (clinical response -100 plus CDAI<150) at week 8 (WOCF).
  Complete remission was defined as CDAI score decrease of ≥100 points from baseline and CDAI score <150 in subjects who had no change in concomitant medications for Crohn's disease except for steroids, which could be tapered after Week 8.
  The CDAI consists of eight variables, including Liquid or very soft stools, Abdominal pain, General well-being, Features of extra-intestinal disease, Oplates for diarrhea, Abdominal mass, Hematocrit and Body weight below standard, each weighted according to its ability to be predictive of disease activity. The total score ranges from 0 to over 600 with higher scores indicating higher disease activity or worse outcome.
Time Frame: 8 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | HMPL-004 | Placebo
Number analyzed (Participants) | 51 | 50
Participants | 13 | 7

12. Secondary Outcome: Complete Remission at Week 12
Description: Percentage of subjects achieving complete remission (clinical response -100 plus CDAI<150) at week 12 (WOCF).
  Complete remission was defined as CDAI score decrease of ≥100 points from baseline and CDAI score <150 in subjects who had no change in concomitant medications for Crohn's disease except for steroids, which could be tapered after Week 8.
  The CDAI consists of eight variables, including Liquid or very soft stools, Abdominal pain, General well-being, Features of extra-intestinal disease, Oplates for diarrhea, Abdominal mass, Hematocrit and Body weight below standard, each weighted according to its ability to be predictive of disease activity. The total score ranges from 0 to over 600 with higher scores indicating higher disease activity or worse outcome.
Time Frame: 12 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | HMPL-004 | Placebo
Number analyzed (Participants) | 51 | 50
Participants | 9 | 5

ADVERSE EVENTS:
Time Frame: From subject randomization through 8 weeks of treatment and through the 30 day follow up period following the date of the last dose of study drug was taken.
Arm/Group | HMPL-004 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 2/51 | 4/50
Other Adverse Events (participants affected / at risk) | 26/51 | 18/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | HMPL-004 (N=51) | Placebo (N=50)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1/28 | 0/29
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Crohn's disease (flare) (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HMPL-004 (N=51) | Placebo (N=50)
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Vomiting (General disorders) | 3 | 2
Pyrexia (General disorders) | 5 | 1
Nasopharyngitis (Infections and infestations) | 5 | 1
Urinary Tract Infection (Infections and infestations) | 3 | 1
Headache (Nervous system disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less